CLINICAL TRIAL: NCT01913964
Title: Acetyl-L-Carnitine Supplementation During HCV Therapy With Pegylated Interferon-α2b Plus Ribavirin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Mariano Malaguarnera, Associate Professor, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10/1997
Record Dates: First submitted 2013-07-26; First posted 2013-08-01 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Work Productivity and Activity Impairment in Workers With Chronic C Hepatitis; Fatigue in Workers With Chronic C Hepatitis; Fatigue
MeSH Terms: conditions — Fatigue | interventions — Acetylcarnitine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetyl-L-carnitine (Experimental): 2 g daily for 12 months
  Interventions: Drug: Acetylcarnitine
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylcarnitine
  Arms: Acetyl-L-carnitine
Drug: Placebo — (sugar pill)
  Arms: placebo

SUMMARY:
To assess the effects of Acetyl-L-Carnitine administration on work productivity, daily activity, and fatigue in subjects with chronic hepatitis C treated with Pegylated-Interferon-α2b and Ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* workers who were 18 years of age or older
* Workers who were infected by HCV and had a quantifiable serum HCV RNA level (as determined by polimerase chain reaction, COBAS AmpliPrep/COBAS TaqMan - ROCHE)
* Cirrhotic workers with a Child-Pugh score less than 7

Exclusion Criteria:

* workers who had other liver diseases
* cancer
* severe jaundice
* pulmonary and renal chronic diseases,
* prostatic diseases
* autoimmune diseases
* diabetes mellitus
* decompensated cirrhosis
* pregnancy
* cardiopathy
* hemoglobinopathies
* hemocromatosis
* major depression
* severe psychiatric pathological conditions

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1997-10; Primary Completion 1997-10 (Actual); Study Completion 1997-10 (Actual)

PRIMARY OUTCOMES:
Work Productivity and Activity Impairment in workers with chronic hepatitis C | 12 months
  Work productivity loss, impairment in daily activities, presenteeism, absenteeism, will be assessed using the Work Productivity and Activity Impairment questionnaire.

SECONDARY OUTCOMES:
Fatigue in workers with chronic hepatitis C | 12 months
  Severity of fatigue, mental fatigue and physical fatigue.